CLINICAL TRIAL: NCT03804905
Title: A Pilot Pragmatic Randomized Controlled Trial to Evaluate the Impact of Improving Access to Drugs on Type 2 Diabetes Care, Outcomes and Costs
Brief Title: STUDIIO-Diabetes Pilot: STUdy of Drug Insurance to Improve Outcomes of Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 103-2018
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus; Medication Adherence; Medication Compliance; Medication Nonadherence
Keywords: Type 2 Diabetes Mellitus; Medication Compliance; Medication Insurance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-cost Medications (Experimental): Eligible patients of physicians allocated to the no-cost medications arm will receive free medications through Trillium Health Partners outpatient pharmacy.
  Interventions: Other: No-cost Medications
- Usual care (No Intervention): Eligible patients of physicians allocated to the usual care arm will continue to access their medications through self-pay or other mechanisms.

INTERVENTIONS:
Other: No-cost Medications — Patients will be connected to Trillium Health Partners outpatient pharmacy, and they will be given an information sheet with further details. The patients will get free access to diabetes, blood pressure and cholesterol medications and for glucose test strips. They can attend the pharmacy in person or arrange for home delivery.
  Arms: No-cost Medications

SUMMARY:
Canada is the only country with a universal health insurance system that does not provide coverage for prescription drugs to all residents. One-third of working-age Canadians have no insurance. Importantly, many of these uninsured patients already face other barriers to good health: low income, new immigrants, single mothers, etc. For these patients, taking prescription drugs - especially chronic disease treatments that may be required lifelong - can be difficult due to high costs. Patients skip doses, delay renewing prescriptions, or simply do not fill prescriptions recommended by their doctors, because they do not have insurance to cover the costs of prescriptions. Previous research by the study team has suggested that the lack of a universal drug insurance program for working-age Canadians affects the health and well-being of low-income people with diabetes. The goal of this research is to determine the clinical and economic impact of providing drug coverage for uninsured type 2 diabetics.

DETAILED DESCRIPTION:
Previous research has found that lowering patients' out-of-pocket costs has a positive impact on health service utilization, risk factor control and patient-reported health for many chronic diseases, including diabetes, hypertension, HIV and asthma. Among patients with chronic disease, medication adherence was inversely associated with hospitalization rates and total healthcare costs, and these relationships were far stronger for diabetes than for any other chronic disease. A recent meta-analysis of eight observational studies showed that adherence with diabetes medications is associated reduction in cardiovascular events, all-cause mortality and all-cause hospitalization. However, virtually all of this previous research has been observational. Only one rigorous intervention study has examined the impact of reducing patient borne drug costs on clinical outcomes. The outcome of this study showed that free medications led to health outcome improvements and a trend towards lower costs.

The goal of this research project is to determine the impact of providing drug coverage to uninsured individuals with one of the most costly chronic diseases, type 2 diabetes. The ultimate goal is to evaluate if lowering out-of-pocket drug costs for uninsured patients is effective and cost-effective to reduce disease morbidity and mortality. Will policy intervention to reduce patients' drug costs would actually translate into improvements in their health outcomes? What impact a universal program would have on overall drug utilization? What total budget impact such a program might have? What extent the cost savings accrued from improving health outcomes might offset the program's implementation costs. Answering these questions will provide essential evidence to inform decision making for a national publicly-funded pharmacare program.

It will demonstrate how medication utilization changes when access improves, and will identify if barriers to utilization other than affordability exist. Crucially, the economic analyses will help policy makers understand the budget impact and cost-effectiveness of a pharmacare intervention. Thus, this research will provide vital information for policy makers crafting a program to provide free drugs to all uninsured Canadians with chronic disease. Such a program is anticipated to have a positive impact on patient experience: to improve health equity and access for vulnerable patients; to facilitate greater medication adherence; and to enhance shared decision-making between patients and their clinicians for effective self-management care paths. The ultimate impact of this research will be evidence for the cost effectiveness or even cost savings of a drug insurance program aimed at the improving access to medications for disadvantaged patients who are currently uninsured.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 2 diabetes record in family physician's electronic medical record
* lack of medication insurance

Exclusion Criteria:

-

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lacking medication insurance | During 2 month run-in period
  Proportion of type 2 diabetes patients aged 25 to 64 who self-report that they lack medication insurance

SECONDARY OUTCOMES:
Online questionnaire during the run-in period | During 2 month run-in period
  Proportion of type 2 diabetes patients aged 25 to 64 who complete the secure online questionnaire during the run-in period
Response to the insurance status question | During 2 month run-in period
  Proportion of type 2 diabetes patients aged 25 to 64 who responded to the insurance status question on the online questionnaire
Recipient of no-cost medications | One year
  Proportion of patients in the intervention group who receive medications from the Trillium Health Partners outpatient pharmacy
Time from allocation to use of Trillium Health Partners outpatient pharmacy | One year
  Time from allocation to the intervention group to use of the Trillium Health Partners outpatient pharmacy

OTHER OUTCOMES:
All-cause mortality or cardiovascular complications | One year
  All-cause mortality, or hospitalization for myocardial infarction, acute coronary syndrome, coronary revascularization, stroke or heart failure.
Other chronic diabetes complications | One year
  Amputation, retinal photocoagulation, vitrectomy, intravitreal injection, incident microalbuminuria, incident chronic kidney disease
Acute diabetes complications | One year
  Emergency department visit or hospitalization for hypo or hyperglycemia
A1c control | One year
  A1c level
Blood pressure control | One year
  Systolic and diastolic blood pressure levels
LDL-cholesterol control | One year
  LDL-cholesterol levels
Medication adherence for study drugs | One year
  Medication possession ratio
Medication adherence for non-study drugs | One year
  Medication possession ratio
Health care utilization | One year
  Ambulatory physician visits, emergency department visits, hospitalizations
Health care costs | One year
  Total health care costs across sectors